CLINICAL TRIAL: NCT05697484
Title: The Impact of Arabic Gamified Mobile Application on Diabetes Control in Egyptian Pediatric Patients With Type 1 Diabetes.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Esmail Alsadek Sherif, Teaching Assistant at faculty of pharmacy, Cairo university, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CL(3017)
Record Dates: First submitted 2023-01-14; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Diabetic Pediatric Patients With Type 1 Diabetes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator)
  Interventions: Device: educational game
- control group (No Intervention)

INTERVENTIONS:
Device: educational game — Control group will be provided with usual care. Intervention group will be provided in addition to the usual care, an access to the mobile game after a simple training for game usage. Both groups will be followed for a period of 3 months.
  The mobile game is planned to have the following design:
  1. Game will be presented in Arabic language.
  2. The game will consist of four levels. a. At the beginning of each level there will be an educational video that the patient must watch in order to be allowed to start the level.
  Arms: intervention group

SUMMARY:
This is a prospective randomized parallel two group pharmacist-led interventional study. The study will involve introduction of the mobile game to pediatric diabetic patients to improve their blood glucose level. The outcomes to be measured are diabetes control and behavioral change in pediatric patients with type1 diabetes mellitus

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients age from 7 to 14 years old to be able to deal with and understand the game.
2. Children previously diagnosed with type1 DM.
3. Arabic speaker.
4. Smart phone (android) access at home, either the mobile of the child or his/her parents.

Exclusion Criteria:

1. Severe cognitive or psychiatric conditions that prevent a patient from understanding the game. any disorder that significantly impairs the cognitive function of an individual to the point where normal functioning in society is impossible without treatment ,examples: dementia- developmental disorders-motor skills disorders- amnesia- substance induced cognitive impairment)25
2. Diabetic pediatric patients at goal with HbA1c < 7.

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
diabetes control | 3 months
  diabetes control that will be assessed by measuring the HbA1c level at baseline and at the end of the study in both groups

SECONDARY OUTCOMES:
Behavioral change | 3 months
  The disease care activities of pediatric diabetic patients will be measured at baseline and at the end of the study after 3 months using The Arabic Summary of Diabetes Self-Care Activities measure.
Measurement of blood glucose control | 3 months
  the random blood glucose level of pediatric patients will be measured by themselves or by their parents on daily basis using glucometer and the reading will be recorded until next visit.
Usability and satisfaction | 3 months
  Usability and satisfaction of the patients will be assessed using a 10-item Arabic System Usability Scale (A-SUS) for mobile applications.

IPD SHARING:
Plan to Share IPD: No